CLINICAL TRIAL: NCT06937931
Title: A Phase II, Multicentre, Randomised, Double-blind, Parallel-Group, Placebo Controlled Study to Evaluate the Efficacy and Safety of IPN10200 as a Treatment for Cervical Dystonia in Adult Participants
Brief Title: A Study of IPN10200 for the Treatment of Cervical Dystonia in Adults
Acronym: CATALPA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLIN-10200-457
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Cervical Dystonia
MeSH Terms: conditions — Torticollis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group 1: Treatment Arm A (Experimental): IPN10200- Dose A
  Interventions: Biological: IPN10200
- Group 1: Treatment Arm B (Experimental): IPN10200- Dose B
  Interventions: Biological: IPN10200
- Group 1: Placebo Comparator (Placebo Comparator): Placebo- Group1
  Interventions: Other: Placebo
- Group 2: Treatment Arm C (Experimental): IPN10200- Dose C
  Interventions: Biological: IPN10200
- Group 2: Placebo Comparator (Placebo Comparator): Placebo- Group 2
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: IPN10200 — Study intervention will be administered in a single treatment cycle after randomisation (Day 1). The administration cycle consists of intramuscular injection.
  Arms: Group 1: Treatment Arm A; Group 1: Treatment Arm B; Group 2: Treatment Arm C
Other: Placebo — Excipients without active substance will be administered in a single treatment cycle after randomisation (Day 1). The administration cycle consists of intramuscular injection.
  Arms: Group 1: Placebo Comparator; Group 2: Placebo Comparator

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of the study drug, IPN10200, and to assess how well it works when compared with placebo in treating Cervical Dystonia (CD) in adults.

CD can cause a series of abnormalities and symptoms in the head and neck that can lead to neck pain and stiffness, and headaches. CD is believed to involve deep parts within the brain that control movement, but genetic factors, environmental factors, and abnormalities in the brain may also play a role.

The usual treatment for CD includes injecting BoNT into the affected muscles, but the treatment only lasts about 3 months. IPN10200 is designed to last for a longer period.

The study will consist of two periods:

1. A Screening Period of up to 4 weeks (28 days) to assess whether a participant can take part in the study and requires at least one visit.
2. A Treatment Period of 36 weeks.

On Day 1 of the treatment period, participants will receive either IPN10200 Dose A or Dose B (additional participants may receive IPN10200 Dose C) of the study drug, or placebo distributed into different muscles in the head, neck and shoulders. Participants may continue some other medications, but details need to be recorded.

There will be 10 visits to the clinic in person and one remote visits (phone call) (12 visits to the clinic for participants who receive Dose C). Participants will undergo blood samplings, urine collections, physical/neurological examinations, and clinical evaluations. Participants will also need to complete questionnaires throughout the study.

The total study duration for a participant will be up to 40 weeks (approximately 9 months).

ELIGIBILITY:
Inclusion Criteria:

1. A clinical diagnosis of isolated Cervical Dystonia (CD) (idiopathic) characterized by dystonic symptoms localised to the head, neck, and shoulder areas with at least moderate severity at Screening and Baseline (Day 1) defined as:

   * (a) Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS)-Total score ≥20
   * (b) TWSTRS-Severity subscale score ≥15
   * (c) TWSTRS-Disability subscale score ≥3
   * (d) TWSTRS-Pain subscale score ≥ 1
2. Treatment naïve or non-naïve to BoNT therapy for CD

Exclusion Criteria:

1. Participants presenting with a swallowing disorder of any origin which might be exacerbated by BoNT treatment, such as:

   * (a) Grade 3 or 4 on the Dysphagia Severity Scale (severe dysphagia) with swallowing difficulties and requiring a change in diet.
2. Predominant anterocollis.
3. Predominant retrocollis.
4. Traumatic torticollis or tardive torticollis.
5. Marked limitation on passive range of motion that suggests cervical contractures or structural abnormality.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2027-03-26 (Estimated); Study Completion 2027-11-05 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) total score | At Week 4
  The Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) is a rating scale for Cervical Dystonia (CD) consisting of three subscales: severity, disability and pain scales. The total score is the sum of each of the subscales, with a range of 0 to 85, where higher scores are indicative of greater impairment.

SECONDARY OUTCOMES:
Change from Baseline in the TWSTRS total score at all other scheduled timepoints post injection until Week 36 | At all timepoints post injection until Week 36.
  The Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) is a rating scale for Cervical Dystonia (CD) consisting of three subscales: severity, disability and pain scales. The total score is the sum of each of the subscales, with a range of 0 to 85, where higher scores are indicative of greater impairment.
Change from Baseline in the TWSTRS-Pain Subscale | At all timepoints post injection until Week 36.
  The TWSTRS pain subscale consists of three patient-rated items that assess the participants usual, worst and best pain from the preceding week, and the subscore has a maximum of 20.
Change from baseline in the daily Numerical Rating Scale (NRS) score | Averaged over every 7-day period until the Week 4 visit
  The Numeric Rating Scale (NRS) is a unidimensional measure of pain intensity in adults. The NRS is a segmented numeric version of the visual analogue scale in which a respondent selects a whole number (0 to 10 integers) that best reflects the intensity of his/her pain. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Time to onset of pain reduction | From study injection to first timepoint at which at least 2-point reduction is observed in NRS score
  Defined as the duration from the administration of the study injection to the first recorded instance of a minimum 2-point decrease in the Numeric Rating Scale (NRS) score.
Time to return of symptoms in responders (time from treatment to loss of 80% of peak treatment effect) | From randomization until Week 36
  As assessed by TWSTRS total score. TWSTRS scale consisting of three subscales: severity, disability and pain scales. The total score is the sum of each of the subscales, with a range of 0 to 85, where higher scores are indicative of greater impairment.
Change from Baseline in the TWSTRS-Disability Subscale | At all timepoints post injection until Week 36.
  The TWSTRS disability subscale assesses the effect that Cervical Dystonia (CD) has on the participant's daily activities and the subscore has a maximum of 30 and consists of six items.
Change from Baseline in the TWSTRS-Severity Subscale | At all scheduled timepoints post injection until Week 36
  The TWSTRS severity subscale rates the maximal excursion of the torticollis (degree of tilt or rotation), elevation, range of motion, etc. This severity subscore has a maximum subtotal of 35 and consists of 11 items.
Change from baseline in Clinical Global Impression of Severity score | At all timepoints post injection until Week 36.
  The Clinical Global Impression of Severity (CGI-S) is a clinician rated scale that measures the severity of an illness in a participant. It is rated on a 7-point scale ranging from 1 (normal) to 7 (severely ill) in answer to a question on the mental state of the participant at the time of the assessment.
Clinical Global Impression of Change score | At all timepoints post injection until Week 36.
  The Clinical Global Impression of Change (CGI-C) is a clinician rated scale that measures the clinical change in a participant. It is rated on a 7 point scale ranging from 1 (very much improved) to 7 (very much worse) in answer to a question on the mental state of the participant at the time of the assessment.
Change from baseline in Patients' Global Impression of Severity score | At all timepoints post injection until Week 36
  The Patient Global Impression of Severity (PGI-S) is a global index that may be used to rate the severity of a specific condition (a single-state scale). The PGI-S is a single question asking the participant to rate how their condition is now on a scale of 1 (Normal) to 4 (Severe).
Patients' Global Impression of Change score | At all timepoints post injection until Week 36
  The Patient Global Impression of Change (PGI-C) is a single-item questionnaire used to measure the participant's impression of overall change in CD, in terms of activity, limitations, symptoms, emotions, and overall quality of life, since the first dose of study intervention. The measure uses a 7-point rating scale with responses ranging from "very much improved" (3) to "very much worse" (-3). Improvement is considered as very much improved, much improved, or minimally improved.
Change from Baseline in the CDIP-58 total score | At all timepoints post injection until Week 36
  The Cervical Dystonia Impact Profile (CDIP-58) is a patient-based rating scale measuring the health impact of CD and contains eight subscales measuring head and neck symptoms (6 items), pain and discomfort (5 items), sleep (4 items), upper limb activities (9 items), walking (9 items), annoyance (8 items), mood (7 items), and psychosocial functioning (10 items). The total score and each subscale score have a common range of 0 (no impact) to 100 (most impact).
Percentage of participants experiencing any Adverse Event (AEs) including treatment emergent adverse events (TEAEs), serious adverse events (SAEs), adverse event of special interest (AESI) and AE leading to treatment discontinuation | From baseline to Week 36.
  An Adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAE is an AE for which the start date is on or after the date that the intervention began.
Percentage of participants with clinically significant changes from baseline in Laboratory Parameters | At all timepoints post injection until Week 36
  Clinically significant change in laboratory parameters will be reported. The clinical significance will graded by the investigator.
Percentage of Participants With Clinically Significant Changes from baseline in Vital Signs | At all timepoints post injection until Week 36
  Clinically significant changes in vital signs will be reported. The clinical significance will be graded by the investigator.
Percentage of participants with clinically significant change from baseline in focused neurological/physical examinations. | At all timepoints post injection until Week 36
Percentage of participants with clinically significant change from baseline in 12-lead Electrocardiogram (ECG) readings. | At all timepoints post injection until Week 36
Treatment-emergence of suicidal ideation/suicidal behaviour | From baseline to Week 36.
  The Columbia Suicide Severity Rating Scale (C-SSRS) will be used in this study for the evaluation of suicidal ideation and behaviour.
Percentage of participants with Binding antibodies to IPN10200 | At all timepoints post injection until Week 36
Percentage of participants with neutralising antibodies to IPN10200 | At all timepoints post injection until Week 36

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (44):
- United States (9):
  - University of Arizona Health Sciences - Neurology, Tucson, Arizona
  - Parkinson's & Mvmt Disorders Inst, Fountain Valley, California
  - Parkinson's Ds & Mvt Disorders Cntr, Boca Raton, Florida
  - USF Health Byrd Alzheimer's Institute, Tampa, Florida
  - Emory Brain Health Center, Atlanta, Georgia
  - Rush Medical Center, Chicago, Illinois
  - Quest Research Institute, Farmington Hills, Michigan
  - Ichan Sch of Medicine @ Mt. Sinai, New York, New York
  - Kingfisher Cooperative, Spokane, Washington
- Czechia (5):
  - Fakultni nemocnice u sv. Anny v Brne - I. Neurologicka klinika, Brno
  - MINKSneuro s.r.o., Brno
  - NEUROHK s.r.o., Choceň
  - Fakultni nemocnice Olomouc - Neurologicka klinika, Olomouc
  - Vseobecna fakultni nemocnice v Praze - Neurologicka klinika, Prague
- France (5):
  - CHU Grenoble Alpes - Site Nord - Neurology, Grenoble
  - Timone University Hospital, Marseille
  - CHU Nimes - Hôpital Caremeau, Nîmes
  - Hopitaux Universitaire de Strasbourg - Hopital de Hautepierre - Neurologie, Strasbourg
  - Centre Hospitalier Universitaire (CHU) Purpan - Institut Des Sciences du Cerveau De Toulouse (Institute for Brain Sciences), Toulouse
- Germany (4):
  - Curiositas ad sanum Studien- und Beratungs GmbH Haag i.OB - Neurologie, Haag in Oberbayern
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - GFO Kliniken Troisdorf, Troisdorf
  - University Hospital Tuebingen - Neurologie, Tübingen
- Italy (5):
  - Ospedale Bellaria, IRCCS Istituto delle Scienze Neurologiche, AUSL Bologna, Bologna
  - Istituto Auxologico Italiano - Auxologico San Luca, Milan
  - Istituto Neurologico C. Besta, Milan
  - IRCCS C.Mondino, Istituto Neurologico Nazionale, Fondazione, Pavia
  - Azienda USL-IRCCS di Reggio Emilia - Presidio ospedaliero provinciale sede di Reggio Emilia, Reggio Emilia
- Poland (7):
  - Specjalistyczna Praktyka Lekarska Dr Stanislaw Ochudlo, Katowice
  - Futuremeds Krakow, Krakow
  - SP ZOZ Szpital Uniwersytecki w Krakowie, Krakow
  - Instytut Zdrowia Dr Boczarska-Jedynak Sp. z o.o. S.K., Oświęcim
  - Eskulap Pabianice Sp z o.o., Pabianice
  - ETG Neuroscience Sp. z o.o., Warsaw
  - Wojewodzki Szpital Specjalistyczny im. J. Gromkowskiego, Wroclaw
- Spain (5):
  - Hospital de la Santa Creu i Sant Pau - Neurología, Barcelona
  - H.U. Puerta del Mar - Neurocirugía, Cadiz
  - Hospital Universitario De La Princesa, Madrid
  - Hospital Universitario Ramon y Cajal - Neurologia, Madrid
  - Hospital Universitario Virgen del Rocio - Neurofisiología Clínica, Seville
- United Kingdom (4):
  - Royal Devon And Exeter Hospital - Neurology, Exeter
  - The Walton Centre, Fazakerley
  - University College London Hospitals NHS Foundation Trust - National Hospital for Neurology and Neurosurgery, London
  - Luton And Dunstable Hospital - Neurology, Luton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and/or EU.
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/